CLINICAL TRIAL: NCT03242148
Title: The Evaluation of the Toffee Nasal Pillows Mask for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: Aspen Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA 219
Record Dates: First submitted 2017-07-25; First posted 2017-08-08 (Actual); Results first posted 2021-06-01 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Toffee Nasal Pillows Mask (Experimental): Participants will be placed on this arm for a total of 14 +- 5 days from visit 2. participants will be using the Toffee mask during this treatment arm
  Interventions: Device: Toffee Nasal Pillows Mask

INTERVENTIONS:
Device: Toffee Nasal Pillows Mask — Participants will be placed on this intervention for a total 14 ± 5 days from Visit 2. Participants will be using the Toffee nasal pillows mask during this treatment arm.

SUMMARY:
This investigation is a prospective, non-randomized, non-blinded study. This investigation is designed to evaluate the performance, comfort and ease of use of the F&P Toffee nasal pillows mask amongst obstructive sleep apnea (OSA) patients. Up to 45 OSA patients will be recruited from the Ohio Sleep Medical Institute (OSMI)

DETAILED DESCRIPTION:
Visit 1 will involve the participants being consented into the trial. Visit 2 will involve the participants being fitted with the F&P Toffee nasal pillows mask for use in-home.

The participant will then come in to return the mask (Visit Three) and have a final interview, this ensures the maximum time participants will be exposed to the Toffee mask in home will be 14 ± 4 days from visit two.

The mask will be returned to the Institution at the conclusion of the trial and the participant will return to their previous mask. The Institution will recruit all patients within 1 week of the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (22+ years of age)
* Able to give informed consent
* Apnea hypopnea Index (AHI) ≥ 5 on diagnostic night
* Either prescribed Automatic positive airway pressure (APAP), Continuous positive airway pressure (CPAP) or Bi-level positive airway pressure (PAP) for OSA
* Fluent in spoken and written English
* Existing nasal pillows mask user

Exclusion Criteria:

* Inability to give informed consent
* Participant intolerant to PAP
* Anatomical or physiological conditions making PAP therapy inappropriate
* Current diagnosis of respiratory disease or carbon Dioxide (CO2) retention
* Pregnant or may think they are pregnant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-09-16 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asim Roy, Principal Investigator — Board Certified Sleep Specialist
Locations (1):
- Ohio Sleep Medicine Institute, Dublin, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Toffee Nasal Pillows Mask
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Toffee Nasal Pillows Mask
Number analyzed (Participants) | 38
Age, Customized [Count of Participants; unit: Participants]
  22-35 | 0
  36-45 | 5
  46-55 | 3
  56-65 | 10
  66-75 | 14
  76-85 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Toffee Mask Usability
Description: Questionnaire on usability during second visit - Subjective.
  Participants rated overall usability of the mask on a 5 point likert type scale ranging from very easy, easy, neither, difficult or very difficult.
Time Frame: 14 ± 5 days in-Home
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Nasal Pillows Mask
Number analyzed (Participants) | 38
Participants
  Rating Very easy or easy | 33
  Rating very difficult or difficult | 1
  Rating Neither | 4

2. Primary Outcome: Toffee Mask Comfort
Description: Determine from questionnaires - Subjective
  Participants rated overall comfort of the mask by indicating on a 5 point likert type scale the degree of comfort they felt. Answer responses ranges from very good, good, neither, poor, or very poor
Time Frame: 14 ± 5 days in-Home
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Nasal Pillows Mask
Number analyzed (Participants) | 38
Participants
  Rated very good or good | 31
  Very poor, poor | 2
  Neither | 5

3. Primary Outcome: Toffee Mask Treatment Performance - Subjective
Description: Determined from questionnaires - Subjective
  Participants rated overall performance of the mask on a 5 point likert type scale with responses including very good, good, neither, poor, or very poor
Time Frame: 14 ± 5 days in-Home
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Nasal Pillows Mask
Number analyzed (Participants) | 38
Participants
  Rated very good or good | 30
  Rated poor or very poor | 4
  Rated neither | 4

4. Primary Outcome: Trial Mask Acceptability
Description: Participant count regarding whether they would continue using the trial mask if given the choice.
Time Frame: 14 ± 5 days in-Home
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Nasal Pillows Mask
Number analyzed (Participants) | 38
Participants
  Yes | 27
  No | 11

5. Secondary Outcome: Toffee Mask Treatment Performance - Objective
Description: Objective data recorded from PAP device - Objective
  Apnea hypopnea index (AHI) data extracted from participants therapy efficacy reports was used to assess this outcome. AHI is a measure of disease severity and is used to evaluate treatment efficacy. Data was reported as a "pass" or "fail" based on the change in AHI from baseline to the intervention. If AHI increased by a clinically significant amount (as reviewed by the PI/study staff) this was marked as a fail.
Time Frame: 14 ± 5 days in-Home
Population: 4 data sets were unavailable for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Nasal Pillows Mask
Number analyzed (Participants) | 34
Participants
  Pass | 34
  Fail | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all participants for 1 year from the date informed consent was obtained.
Arm/Group | Toffee Nasal Pillows Mask
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 8/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toffee Nasal Pillows Mask (N=38)
Nasal Irritation (Skin and subcutaneous tissue disorders) | 7 (7)
Sore on the top of the head (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT03242148/Prot_SAP_001.pdf